CLINICAL TRIAL: NCT02252133
Title: Pilot Evaluation of DAILIES TOTAL1® Lens Centration in a Japanese Population
Brief Title: DAILIES TOTAL1® Lens Centration in a Japanese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ALJ-V2014-1
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-11

CONDITIONS: Myopia; Refractive Error
Keywords: Contact lenses; Myopia
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DT1, then 1DAVTE (Other): Delefilcon A contact lenses worn first, followed by narafilcon A contact lenses. Each product worn bilaterally for 7 days on a daily wear, daily disposable basis.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses
- 1DAVTE, then DT1 (Other): Narafilcon A contact lenses worn first, followed by delefilcon A contact lenses. Each product worn bilaterally for 7 days on a daily wear, daily disposable basis.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Silicone hydrogel contact lenses (8.5 and 8.8 base curves) dispensed per manufacturer's guidelines for daily disposable wear
  Other Names: DAILIES TOTAL1®
Device: Narafilcon A contact lenses — Silicone hydrogel contact lenses (8.5 and 9.0 base curves) dispensed per manufacturer's guidelines for daily disposable wear
  Other Names: 1-DAY ACUVUE® TruEye®

SUMMARY:
The purpose of this study is to compare the lens centration of DAILIES TOTAL1® (DT1) contact lenses to 1-DAY ACUVUE® Tru-Eye® (1DAVTE) contact lenses in a Japanese population after 7 ± 2 days of wearing of each product.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Habitually wear soft contact lenses on a daily disposable or weekly/monthly replacement basis.
* Symptoms of contact lens discomfort as defined by protocol.
* Require contact lenses within the power range of -0.50 diopter (D) to -10.00 D.
* Cylinder, if present, less or equal to 0.75D in either eyes at Visit 1.
* Vision correctable to 20/25 or 0.1 (logMAR) or better in each eye at distance with pre-study lenses at Visit 1.
* Acceptable contact lens fit with both study contact lenses.
* Willing to wear lenses every day for at least for a minimum of five days per week six hours per day, every day if possible and attend all study visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing DT1 or 1DAVTE.
* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear.
* Use of systemic or ocular medications which contact lens wear could be contraindicated as determined by the investigator.
* Eye injury or surgery within twelve weeks immediately prior to enrollment for this trial.
* Any moderate or severe ocular condition observed during the slit-lamp examination at the enrollment visit.
* History of herpetic keratitis, ocular surgery or irregular cornea.
* Prior refractive surgery (e.g. LASIK, PRK, etc).
* Monocular subjects (only one eye with functional vision) or subjects fit with only one lens.
* Judged ineligible as a patient in this clinical study by the investigator.
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Clinical Development, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon Japan Ltd. for Trial Locations, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 study centers located in Japan.
Pre-assignment Details: Of the 53 enrolled, 6 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (47).
Period: Period 1
Arm/Group | DT1, Then 1DAVTE | 1DAVTE, Then DT1
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Period 2
Arm/Group | DT1, Then 1DAVTE | 1DAVTE, Then DT1
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized subjects.
Groups:
- Overall: DAILIES TOTAL1® and 1-Day Acuvue® TruEye® contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Lens Centration After 7 ± 2 Days of Wear
Description: Lens centration (the centration of the contact lens over the cornea) was rated by the investigator during slit lamp examination using a 5-point scale (0=optimal, 4=severe decentration). Success was defined as the percentage of subjects whose lens centration was rated as "optimal" or "slight decentration. One eye (study eye) was analyzed.
Time Frame: Day 7, each product
Population: This analysis population includes all subjects who used the study lenses and who met all inclusion criteria and did not meet any exclusion criteria.
Measure: Number; unit: percentage of subjects
Groups:
- Dailies Total 1: Delefilcon A contact lenses during Period 1 or Period 2 for 7 days.
- 1DAVTE: Narafilcon A contact lenses worn during Period 1 or Period 2 for 7 days.
Arm/Group | Dailies Total 1 | 1DAVTE
Number analyzed (Participants) | 42 | 45
percentage of subjects | 100.0 | 86.7

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 14 days). AEs were obtained through use of a subjective questionnaire.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device.
Groups:
- Dailies Total 1: All subjects who wore delefilcon A contact lenses
- 1DAVTE: All subjects who wore narafilcon A contact lenses
Arm/Group | Dailies Total 1 | 1DAVTE
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.